CLINICAL TRIAL: NCT00179595
Title: Does the Relaxation Response Inhibit Acute Stress?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2001P001747; H75-CCH-123424; H75-CCH-119124
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Healthy
Keywords: nitric oxide, volumetric oxygen consumption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: relaxation response- meditation

SUMMARY:
The purposes of this study are:

1. To examine molecular and biochemical changes, associated with the relaxation response (RR) that can counteract the effects of stress in healthy adults.
2. To compare genomic, molecular and biochemical parameters between healthy adults with a long term meditative practice and those with no experience in meditation.

Since stress is a factor in the development of many health conditions, a further understanding of the mechanisms of the RR should be developed. The project is designed to determine how the RR can improve the quality of life that has been adversely affected by stress.

DETAILED DESCRIPTION:
The purposes of this study are:

1. To examine molecular and biochemical changes, associated with the relaxation response (RR) that can counteract the effects of stress in healthy adults.
2. To compare genomic, molecular and biochemical parameters between healthy adults with a long term meditative practice and those with no experience in meditation.

Since stress is a factor in the development of many health conditions, a further understanding of the mechanisms of the RR should be developed. The project is designed to determine how the RR can improve the quality of life that has been adversely affected by stress.

ELIGIBILITY:
Inclusion Criteria:

* healthy individual
* age:18-49 years
* able to read and understand English
* able to attend al study visits
* access to a telephone (to schedule visits)

Exclusion Criteria:

* current smoking
* asthma
* current use of any prescription or psychoactive medications or supplements
* either:

  1. no prior experience with RR eliciting techniques
  2. at least 3 years of regular RR elicitation (at least 20 min/day)
* BMI >30
* exhaled nitric oxide levels >60 ppb
* abnormal lab values (Hct <32,creatinine >1.3, glucose >200
* pregnancy

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2002-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To examine molecular and biochemical changes, associated with the relaxation response (RR) that can counteract the effects of stress in healthy adults.

SECONDARY OUTCOMES:
To compare genomic, molecular and biochemical parameters between healthy adults with a long term meditative practice and those with no experience in meditation.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Benson, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth-Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No